CLINICAL TRIAL: NCT06075953
Title: DCIS: RECAST Trial -Ductal Carcinoma In Situ: Re-Evaluating Conditions for Active Surveillance Suitability as Treatment: a Breast Cancer Prevention Pilot Study
Brief Title: DCIS: RECAST Trial Ductal Carcinoma In Situ: Re-Evaluating Conditions for Active Surveillance Suitability as Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QuantumLeap Healthcare Collaborative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECAST-DCIS
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ductal Carcinoma in Situ
Keywords: active surveillance; hormone therapy; endocrine therapy
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Tamoxifen; exemestane; Letrozole; Anastrozole; Testosterone; elacestrant; 4-hydroxy-N-desmethyltamoxifen

STUDY DESIGN:
Intervention Model Description: RECAST-DCIS is an open-label, multi-site platform study designed to offer women with Ductal cell Carcinoma In Situ (DCIS) 6 months of neo-adjuvant exposure to endocrine therapy with the intent of determining their suitability for long-term active surveillance without surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- chemoprevention therapy per investigator choice (Active Comparator): For premenopausal women: 20 mg tamoxifen orally daily (standard dose) or 10 mg every other day (low dose).
  For postmenopausal women: standard oral doses of AI of choice: exemestane 25 mg daily, letrozole 2.5 mg daily, or anastrozole 1 mg daily; or reduced exemestane dosing: 25 mg 3X per week orally.
  For postmenopausal women who are not tolerating an AI, investigators can change them to the low dose (10 mg every other day) or standard dose (20 mg) of tamoxifen.
  There is active follow up with MRI at baseline, 3 months, 6 months after treatment initiation, and every 6 months alternating MRI and mammogram for up to 5 years. Participants may continue treatment for up to 5 years.
  Interventions: Drug: Tamoxifen; Drug: Exemestane; Drug: Letrozole; Drug: Anastrazole
- Testosterone + Anastrazole (T+Ai) (Experimental): White solid pellet for subcutaneous insertion consisting of 100mg Testosterone and 4mg Anastrazole, an aromatase inhibitor. A cylindrical pellet (4.5mm diameter, 6.35mm diameter) is inserted subcutaneously in the upper outer gluteal region or iliac fossa every 3 months, with treatment up to 36 months. There is active follow up with MRI at baseline, 3 months, 6 months after treatment initiation, and every 6 months alternating MRI and mammogram for up to 5 years. Participants are followed for an additional 5 years.
  Interventions: Drug: Testosterone + Anastrazole
- Elacestrant (Experimental): Selective estrogen receptor degrader, Standard dose: 400mg PO with food once daily for treatment up to 36 months. Dose reduction of Elacestrant by up to 2 dose levels permitted depending on toxicity; 400 mg to 300 mg then 300 mg to 200 mg Participants requiring more than 2 dose reductions must discontinue treatment For patients on this arm there is active follow up with MRI at baseline, 3 months, 6 months after treatment initiation, and every 6 months alternating MRI and mammogram for up to 5 years. Participants are followed by for an additional 5 years.
  Interventions: Drug: Elacestrant
- Endoxifen (Experimental): (Z)-endoxifen is the most active metabolite of the selective estrogen receptor modulator (SERM), tamoxifen. Standard dose: 10mg PO delayed release capsule of z-endoxifen once daily for treatment up to 36 months. same time with a glass of water either 1 hour before a meal or 2 hours after a meal and should not take with alcohol. For patients on this arm there is active follow up with MRI at baseline, 3 months, 6 months after treatment initiation, and every 6 months alternating MRI and mammogram for up to 5 years. Participants are followed for an additional 5 years.
  Interventions: Drug: Z-endoxifen

INTERVENTIONS:
Drug: Tamoxifen — For premenopausal women: 20 mg tamoxifen orally daily (standard dose) or 10 mg every other day (low dose).
  For postmenopausal women who are not tolerating an AI, investigators can change them to the low dose (10 mg every other day) or standard dose (20 mg) of tamoxifen.
  Arms: chemoprevention therapy per investigator choice
Drug: Exemestane — For postmenopausal women: standard oral doses of AI of choice: exemestane 25 mg daily, or reduced exemestane dosing: 25 mg 3 times per week orally
  Arms: chemoprevention therapy per investigator choice
Drug: Letrozole — For postmenopausal women: standard oral doses of AI of choice: letrozole 2.5 mg daily.
  Arms: chemoprevention therapy per investigator choice
Drug: Anastrazole — For postmenopausal women: standard oral doses of AI of choice: anastrozole 1 mg daily.
  Arms: chemoprevention therapy per investigator choice
Drug: Testosterone + Anastrazole — Investigational drug. Both pre- and post- menopausal subjects. 100mg testosterone in combination with 4mg anastrazole administered subcutaneously every 3 months for up to 3 years.
  Other Names: T+Ai
  Arms: Testosterone + Anastrazole (T+Ai)
Drug: Elacestrant — Investigational drug. Both pre- and post- menopausal subjects. Elacestrant 400mg PO with food once daily up to 36 months.
  Arms: Elacestrant
Drug: Z-endoxifen — Investigational drug. Both pre- and post- menopausal subjects. (z)-endoxifen 10mg delayed release capsule 1 hour before a meal or 2 hours after a meal once daily for up to 36 months.
  Arms: Endoxifen

SUMMARY:
The goal of this trial is to see if active surveillance monitoring and hormonal therapy in patients diagnosed with ductal cell carcinoma in situ (DCIS), an early stage of breast cancer, can be an effective management of the disease.

Participants will be asked to receive control hormonal therapy or an investigational hormonal therapy treatment. Participants will be asked to return for evaluation with MRI at three months and six months. Depending on the evaluation participants will have the option to continue on the treatment. If the evaluation suggests surgery is recommended, the participant will discontinue the study treatment and will undergo surgery. In addition to the treatment and MRI evaluation, participants will be asked to provide blood sample to understand their immune status, provide saliva sample for genetic testing, provide the study with a portion of the tissue or slides generated from tissue removed during surgery performed as part of their standard of care.

DETAILED DESCRIPTION:
The goal of this trial is to see if active surveillance monitoring and hormonal therapy in patients diagnosed with Ductal cell Carcinoma In Situ (DCIS), an early stage of breast cancer, can be an effective management of the disease. The current management of most patients with DCIS involves surgical intervention with or without radiation, similar to more aggressive breast cancers. These treatments can come with some significant health effects.The main question this study aims to answer is: to determine whether novel endocrine therapy increases the fraction of patients who will be suitable for long-term active surveillance.

Participants will be asked to take one of three investigational study medication (z-Elacestrant, Testosterone + Anastrazole, or Endoxifen) or receive control hormonal therapy (Tamoxifen or an aromatase inhibitor), depending on the treatment to which they have been randomized. Participants will be asked to return for evaluation with MRI at three months and six months. Depending on the evaluation, participants will have the option to continue on the treatment, with follow up evaluations of Mammogram and MRI at 6 month intervals. If the evaluation suggests surgery is recommended, the participant will discontinue the study treatment and will undergo surgery. In addition to the treatment and MRI evaluation, participants will be asked to:

* Provide blood sample to understand their immune status
* Provide saliva sample for genetic testing
* Provide the study with a portion of the tissue or slides generated from tissue removed during surgery performed as part of their standard of care.

Participants will be followed annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

A. Female, at least 18 years old

B. Previous diagnosis of HR+ DCIS (at least 50% ER or PR; biopsy will have been performed previously at diagnosis) with or without microinvasion

C. Patients who have previously received endocrine therapy should have a washout period of 4-6 weeks prior to the screening MRI on the RECAST-DCIS trial

D. Bilateral mammogram performed within up to 4 months (120 days) of the start of trial treatment may be used for screening evaluation

E. MRI performed within up to 2 months (60 days) of the start of trial treatment for lesion evaluation

F. CBC w/ diff, CMP, and Lipid Panel within normal limits within a year of the start of trial treatment. Abnormal labs to be repeated within 60 days prior to the start of trial treatment. Patients will be considered eligible for screening labs that are abnormal or out-of-range if the investigator has deemed the lab results not-clinically significant

G. Negative urine or serum pregnancy test within 1 month of the start of trial treatment

H. Controlled HIV positive patients are allowed as long as their current medication does not contraindicate the study's investigational agent

I. Willingness and ability to provide tumor samples for research

Exclusion Criteria:

A. Pregnant or actively breastfeeding women

B. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent based on review of the medical record and patient history

C. Invasive carcinoma or identification of a mass on MRI that is subsequently biopsied and found to be invasive cancer

D. Co-enrollment in clinical trials of pharmacologic agents requiring an IND

E. Ongoing treatment for DCIS other than what is specified in this protocol

F. Uncontrolled intercurrent illness, including psychiatric conditions, that would limit compliance with study requirements

G. Medical history or ongoing gastrointestinal disorders potentially affecting the absorption of investigational agent and/or tamoxifen. Active inflammatory bowel disease or chronic diarrhea, known active hepatitis A/B/C*, hepatic cirrhosis, short bowel syndrome, or any upper gastrointestinal surgery including gastric resection or banding procedures

*Active hepatitis, defined as: A (positive HA antigen or positive IgM); B (either positive HBs antigen or positive hepatitis B viral DNA test above the lower limit of detection of the assay); C (positive hepatitis C antibody result, and quantitative hepatitis C (HCV) ribonucleic acid (RNA) results greater than the lower limits of detection of the assay)

H. Participants who are unable to swallow normally or unable to take tablets and capsules. Predictable poor compliance with oral treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 400 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Patients remaining on active surveillance at 7 months | 7 months
  Fraction of patients remaining on active surveillance at 7 months compared to control

SECONDARY OUTCOMES:
To determine whether novel endocrine therapy increases the fraction of patients who will be suitable for long-term active surveillance as measured by the fraction of patients deemed to be low-risk for invasive cancer at 6 months compared to control | 6 months
  Fraction of patients categorized as low risk by MRI after 6 months of treatment--Measured by cases demonstrating endocrine responsiveness (Determined based on lesion and background or lesion alone or lack of lesion and minimal background)
To determine whether novel endocrine therapy increases the fraction of patients who will be suitable for long-term active surveillance as measured by the fraction of patients deemed to be low-risk for invasive cancer at 3 months compared to control | 3 months
  Fraction of patients categorized as low risk by MRI after 3 months of treatment--Measured by cases demonstrating endocrine responsiveness (Determined based on lesion and background or lesion alone or lack of lesion and minimal background)
Associate rate of progression to Invasive Ductal Carcinoma (IDC) with risk categorization after 6 months of treatment at 3 years | 3 years
  Correlation of low-risk categorization at 6 months with subsequent rate of Invasive Ductal Cell Carcinoma progression at 3 years
To assess the QoL impact of novel endocrine therapy compared to tamoxifen or Aromatase inhibitor (Ai) at standard or low dose using PROMIS and the FACT-ES and FACT-GP5 composite score compared to control | 6 months
  Fraction of patients experiencing Minimum Important Difference in overall QOL measured by PROP-R statistics (PROMIS) and FACT-ES (functional assessment of cancer therapy- endocrine symptoms) and FACT-GP5, a quality of life (QoL) assessment)
For those with an identified lesion on MRI imaging, determine whether neoadjuvant endocrine therapy decreases lesion volume (qualitative, quantitative) and whether that corresponds to the biologic type of Ductal cell carcinoma In Situ (DCIS) | 6 months
  Rate of reduction in focal lesions (mass and non-mass enhancement (NME) at 6 months and Rate of reduction in focal lesions using automated Functional Tumor Volume
To determine whether neoadjuvant endocrine therapy decreases automated background parenchymal enhancement (BPE and automated MRI density compared to Ai and Tamoxifen | 6 months
  % with contralateral reduction in qualitative and automated BPE and % reduction in contralateral breast density
Determine adherence to active surveillance protocol | 5 years
  Time to discontinuation of therapy (Tolerability of therapy) will be measured, and Adherence rates on each regimen, as well as PROP-R, FACT-ES and FACT-GP5 score on each regimen will be measured. These assessments will be combined to evaluate efficacy and toxicity using a novel clinical benefit index.
Change in artificial intelligence predicted risk based on mammography | 5 years
  Correlation of BPE change with agent and compare to quantitative imaging density

OTHER OUTCOMES:
Assess Germ Line polygenic risk: assess correlation of detectable mutations with endocrine response and qualification for active surveillance at 7 months | 7 months
  evaluate influence of polygenic risk on endocrine response and suitability for Active Surveillance
To evaluate outcomes stratified by immune and molecular subtype based upon multiplex immuno histochemistry (IHC) clustering analysis, and RPS expression array profiling | 7 months
  Response stratified by multiplex immune staining for Human Epidermal growth factor receptor-2 (HER2) isoforms and Response Predictive Subtypes (RPS)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Esserman, MD, MBA, Principal Investigator — University of California, San Fancisco - Department of Surgery; (Co-PI) Kelly Hewitt, MD, FACS, Principal Investigator — Huntsman Cancer Institute at the University of Utah
Locations (26):
- United States (26):
  - Berkeley Outpatient Center, Berkeley, California
  - City of Hope -Duarte Cancer Center, Duarte, California
  - City of Hope - Lennar Foundation Cancer Center, Irvine, California
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - City of Hope, South Pasadena, California
  - John Muir Health, Walnut Creek, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Maple Grove Cancer Center, Maple Grove, Minnesota
  - Hennepin Healthcare -Minneapolis, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Health Partners - Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Health Partners - Regions Hospital, Saint Paul, Minnesota
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No